CLINICAL TRIAL: NCT02190162
Title: A Prospective Double-blined Randomized Trial to Evaluate The Influence of Tantum Verde® on Recovery Following Tonsillectomy
Brief Title: The Influence of Tantum Verde® on Recovery Following Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Ronen Ohad, MD, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0028-14-NHR
Record Dates: First submitted 2014-06-16; First posted 2014-07-15 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Tonsillectomy; Adenoidectomy
Keywords: Patients undergoing tonsillectomy with or without adenoidectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tantum Verde® mouthwash (Active Comparator): solution of Tantum Verde
  Interventions: Drug: Tantum Verde® mouthwash
- placebo mouthwash (Placebo Comparator): saline with mint flavor
  Interventions: Other: Placebo mouthwash

INTERVENTIONS:
Drug: Tantum Verde® mouthwash
  Arms: Tantum Verde® mouthwash
Other: Placebo mouthwash — Mouthwash with placebo solution
  Arms: placebo mouthwash

SUMMARY:
The purpose of this study is to assess the effects of Tantum Verde® for improving recovery following tonsillectomy Study design: A prospective double-blined randomized trial. Sample size: Thirty patients undergoing tonsillectomy who will be treated with Tantum Verde® Mouth wash solution, and a control group of 30 patients that will undergo tonsillectomy and will be treated with a placebo.

The study will be conducted in the Departments Otolaryngology - Head and Neck Surgery in the Western Galilee Medical Center, Nahariya, Israel. Patients who are scheduled for tonsillectomy with or without adenoidectomy will be recruited for the study. They will sign the inform consent in one of two places: in the departments before the surgery or in the clinic in the visit before the surgery. The patients will be evaluated for their ability to gargle and spit water before the surgery, after which they will be assigned to either the treatment group who will get a solution of Tantum Verde or the control group who will receive saline with mint flavor, both in identicle bottles. Randomization will be done using a random number generator program.

The patients will be asked to gargle and spit the solution they received three times a day for 30 seconds, for the following week after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing tonsillectomy with or without adenoidectomy
* Over 12 years of age
* Signed informed consent by patient or caregiver

Exclusion Criteria:

* Inability to gargle and spit
* Allergy to one of the solution ingredients
* Significant comorbidity (e.g. diabetes, bleeding disorders)
* Unable/ unwilling to comply with the protocol requirements
* Pregnancy or breast feeding
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study

Withdrawal Criteria:

• Patients did not comply with the protocol requirements

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Pain: reduction in severity based on VAS score. | postoperative pain using VAS(Visual Analogue Scale) on day 14
Pain: time to complete resolution based on VAS score. | postoperative pain using VAS(Visual Analogue Scale) on day 14
Pain medication: postoperative pain medication type, dosage and reduction in the demand postoperatively | Data of Pain medication: postoperative pain medication type, dosage and reduction in the demand postoperatively will be collected on day 14
Bleeding: time to complete cessation, need for re-operation | bleeding score will be Measured according to:bleeding, no bleeding and surgery required for 14 days after surgery.
Bleeding: postoperative measures to reduce bleeding | bleeding score will be Measured according to:bleeding, no bleeding and surgery required for 14 days after surgery.

SECONDARY OUTCOMES:
Readmission for any reason. | 14 Days after surgery
Duration of hospital stay | day14
Time to return to normal diet and activities. | day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Galillee medical center, Nahariya, Israel